CLINICAL TRIAL: NCT06721975
Title: Prospective Single-center Study Comparing Thulium Fiber Laser to Pulsed Thulium:YAG Laser in the Ureteroscopic Treatment of Nephrolithiasis
Brief Title: Thulium Fiber Laser (TFL) vs Thulio Pulsed Thulium:YAG (p-Tm:YAG)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Dornier MedTech Systems (Industry)
Responsible Party: Principal Investigator, Roger L Sur, M.D., Professor of Urology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 810115; 314954-00001 (Other Grant/Funding Number: Dornier MedTech)
Record Dates: First submitted 2024-11-25; First posted 2024-12-06 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Kidney Stones; Nephrolithiasis
Keywords: laser lithotripsy; laser; nephrolithiasis; kidney stone
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: Patient will be randomized to one of the following two groups:
  1. p-Tm:YAG laser system
  2. TFL laser system
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- p-Tm:YAG laser system (Experimental): This is a new laser system developed by Dornier, the Thulio pulsed Thulium:YAG (p-Tm:YAG)
  Interventions: Device: Thulio pulsed Thulium:YAG (p-Tm:YAG)
- TFL laser system (Active Comparator): The thulium fiber laser (TFL) has demonstrated effectiveness in this procedure.
  Interventions: Device: Thulium Laser Fiber (TFL)

INTERVENTIONS:
Device: Thulio pulsed Thulium:YAG (p-Tm:YAG) — A new laser system developed by Dornier, the Thulio pulsed Thulium:YAG (p-Tm:YAG ) is beginning to be studied in vitro and in vivo. Dornier Thulio p-Tm:YAG may represent an attractive new laser platform, with comparable properties to TFL including decreased retropulsion, smaller dust, and improved ablation efficiency relative to Ho:YAG.
  Arms: p-Tm:YAG laser system
Device: Thulium Laser Fiber (TFL) — The thulium fiber laser (TFL) has demonstrated effectiveness in this procedure
  Arms: TFL laser system

SUMMARY:
This research study is being conducted to assess the ability and efficiency of two laser systems to break up kidney stones during ureteroscopy with laser lithotripsy for kidney stone treatment.

DETAILED DESCRIPTION:
Ureteroscopic stone treatment is a minimally invasive procedure commonly performed for kidney stones. Recently, the thulium fiber laser (TFL) has demonstrated effectiveness in this procedure. A new laser system developed by Dornier, the Thulio pulsed Thulium:YAG (p-Tm:YAG ) is beginning to be studied in vitro and in vivo. Dornier Thulio p-Tm:YAG may represent an attractive new laser platform, with comparable properties to TFL including decreased retropulsion, smaller dust, and improved ablation efficiency relative to Ho:YAG. Moreover, the p-Tm:YAG laser has been shown to be effective in treating a wide range of human stone types. The Dornier Thulio p-Tm:YAG laser has been tested clinically in a limited fashion via pilot studies in URS and the RevoLix Hybrid Thulium Laset (HTL) was studied in mini-PCNL. However, limited research has directly compared its efficacy and safety and no prospective comparative trials have been published.

This study aims to investigate whether Dornier Thulio p-Tm:YAG laser is non-inferior to TFL in terms of dusting ablation efficiency (J/mm3) and dusting ablation speed (mm3/s) for ureteroscopic stone treatment. To our knowledge no large-scale study has examined the outcomes of p-Tm:YAG compared to TFL for the treatment of kidney stones which warrants an investigation giving the promising results previously reported.

The primary objective is to assess stone dusting ablation efficiency (Joules/stone volume ablated) between both laser systems in vivo for ureteroscopic stone treatment . Secondary objectives include assessing stone dusting ablation speed (stone volume ablated/lasing time) and complication profile of both laser systems.

The investigators hypothesize that dusting ablation efficiency and speed of the p-Tm:YAG laser will be non-inferior to TFL for the treatment of renal stones totaling 7-20 mm in diameter with similar clinical and safety/complication outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Solitary renal stone 7 to 20 mm in size or in the case of multiple stones the conglomerate diameter (additive maximal diameter of all stones on axial imaging of computed tomography) of 7-20 mm is required
* Must be a suitable operative candidate for flexible ureteroscopy per American Urological Association guidelines
* Must be able to give consent
* Bilateral ureteroscopy will be permitted but only the first side (per surgeon discretion) will be included in the study
* Surgeons participating in the study must be urological attending surgeons or fellows with subspecialty training in Endourology

Exclusion Criteria:

* Concomitant stones in the ureter
* Prior ipsilateral upper urinary tract reconstructive procedures or history of ipsilateral ureteral stricture
* Prior radiotherapy to the abdomen or pelvis
* Neurogenic bladder or spinal cord injury
* Pregnancy
* Untreated UTI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The amount of energy used per given stone volume | From enrollment to the follow up imaging at 6-12 weeks
  The primary object is to assess the stone dusting ablation efficiency - efficiency will be defined by amount of laser energy used per stone volume (Joules/mm3)

SECONDARY OUTCOMES:
Laser ablation speed (volume of stone/lasing time = mm3/sec) | From enrollment to the follow up imaging at 6-12 weeks
  Secondary objectives include assessing stone dusting ablation speed. This is assessed by taking the stone volume ablated (mm3) and dividing it by lasing time (seconds) - mm3/sec.
Post-operative complications compared between the two laser systems | From enrollment to the follow up imaging at 6-12 weeks
  Secondary objectives include assessing post-operative complications. This is defined as the proportion of post-operative infections, readmissions to the hospital, and unplanned procedures compared between the two laser systems.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wan X, Wang W, Liu J, Tong T. Estimating the sample mean and standard deviation from the sample size, median, range and/or interquartile range. BMC Med Res Methodol. 2014 Dec 19;14:135. doi: 10.1186/1471-2288-14-135. PMID 25524443
- [Background] Ventimiglia E, Robesti D, Bevilacqua L, Tondelli E, Oliva I, Orecchia L, Juliebo-Jones P, Pietropaolo A, De Coninck V, Esperto F, Tailly T, Ferretti S, Gauhar V, Somani B, Villa L, Keller EX, Salonia A, Traxer O, Kartalas Goumas I. What to expect from the novel pulsed thulium:YAG laser? A systematic review of endourological applications. World J Urol. 2023 Nov;41(11):3301-3308. doi: 10.1007/s00345-023-04580-z. Epub 2023 Sep 8. PMID 37682286
- [Background] Ventimiglia E, Pauchard F, Gorgen ARH, Panthier F, Doizi S, Traxer O. How do we assess the efficacy of Ho:YAG low-power laser lithotripsy for the treatment of upper tract urinary stones? Introducing the Joules/mm3 and laser activity concepts. World J Urol. 2021 Mar;39(3):891-896. doi: 10.1007/s00345-020-03241-9. Epub 2020 May 27. PMID 32462304
- [Background] Vaddi CM, Ramakrishna P, Ganeshan S, Swamy S, Anandan H, Babu M, Panda R. The clinical efficiency and safety of 60W superpulse thulium fiber laser in retrograde intrarenal surgery. Indian J Urol. 2022 Jul-Sep;38(3):191-196. doi: 10.4103/iju.iju_60_22. Epub 2022 Jul 1. PMID 35983111
- [Background] Taratkin M, Azilgareeva C, Korolev D, Barghouthy Y, Tsarichenko D, Akopyan G, Chinenov D, Ali S, Kozlov V, Mikhailov V, Enikeev D. Prospective Single-Center Study of SuperPulsed Thulium Fiber Laser in Retrograde Intrarenal Surgery: Initial Clinical Data. Urol Int. 2022;106(4):404-410. doi: 10.1159/000516933. Epub 2021 Jun 16. PMID 34134117
- [Background] Stern KL, Borgert BJ, Wolf JS Jr. Steerable Ureteroscopic Renal Evacuation (SURE) for Large Renal Stones: A Multi-Institutional Center Study. J Endourol. 2023 Aug 28;37(11):1179-83. doi: 10.1089/end.2023.0424. Online ahead of print. PMID 37639362
- [Background] Solano C, Corrales M, Panthier F, Candela L, Doizi S, Traxer O. Navigating urolithiasis treatment: assessing the practicality and performance of thulium fiber laser, holmium YAG, and thulium YAG in real-world scenarios. World J Urol. 2023 Oct;41(10):2627-2636. doi: 10.1007/s00345-023-04487-9. Epub 2023 Jul 20. PMID 37468656
- [Background] Sierra A, Corrales M, Kolvatzis M, Traxer O. Initial clinical experience with the thulium fiber laser from Quanta System: First 50 reported cases. World J Urol. 2022 Oct;40(10):2549-2553. doi: 10.1007/s00345-022-04096-y. Epub 2022 Jul 21. PMID 35861860
- [Background] Petzold R, Suarez-Ibarrola R, Miernik A. Temperature Assessment of a Novel Pulsed Thulium Solid-State Laser Compared with a Holmium:Yttrium-Aluminum-Garnet Laser. J Endourol. 2021 Jun;35(6):853-859. doi: 10.1089/end.2020.0803. Epub 2020 Dec 3. PMID 33191783
- [Background] Petzold R, Suarez-Ibarrola R, Miernik A. Gas Bubble Anatomy During Laser Lithotripsy: An Experimental In Vitro Study of a Pulsed Solid-State Tm:YAG and Ho:YAG Device. J Endourol. 2021 Jul;35(7):1051-1057. doi: 10.1089/end.2020.0526. Epub 2020 Dec 22. PMID 33207950
- [Background] Petzold R, Miernik A, Suarez-Ibarrola R. Retropulsion force in laser lithotripsy-an in vitro study comparing a Holmium device to a novel pulsed solid-state Thulium laser. World J Urol. 2021 Sep;39(9):3651-3656. doi: 10.1007/s00345-021-03668-8. Epub 2021 Mar 23. PMID 33758959
- [Background] Petzold R, Miernik A, Suarez-Ibarrola R. In Vitro Dusting Performance of a New Solid State Thulium Laser Compared to Holmium Laser Lithotripsy. J Endourol. 2021 Feb;35(2):221-225. doi: 10.1089/end.2020.0525. Epub 2020 Sep 9. PMID 32799650
- [Background] Patil A, Reddy N, Shah D, Singh A, Ganpule A, Sabnis R, Desai M. High-Power Holmium with MOSES Technology or Thulium Fiber Laser in MiniPerc with Suction: A New Curiosity. J Endourol. 2022 Oct;36(10):1348-1354. doi: 10.1089/end.2021.0915. Epub 2022 Aug 17. PMID 35331003
- [Background] Panthier F, Solano C, Chicaud M, Kutchukian S, Candela L, Doizi S, Corrales M, Traxer O. Initial clinical experience with the pulsed solid-state thulium YAG laser from Dornier during RIRS: first 25 cases. World J Urol. 2023 Aug;41(8):2119-2125. doi: 10.1007/s00345-023-04501-0. Epub 2023 Jul 6. PMID 37414942
- [Background] Negida A. Sample Size Calculation Guide - Part 6: How to calculate the sample size for a non-inferiority or an equivalence clinical trial. Adv J Emerg Med. 2019 Nov 27;4(1):e15. doi: 10.22114/ajem.v0i0.302. eCollection 2020 Winter. No abstract available. PMID 31938784
- [Background] Kwok JL, Ventimiglia E, De Coninck V, Corrales M, Sierra A, Panthier F, Pauchard F, Schmid F, Hunziker M, Poyet C, Daudon M, Traxer O, Eberli D, Keller EX. Pulsed thulium:YAG laser-ready to dust all urinary stone composition types? Results from a PEARLS analysis. World J Urol. 2023 Oct;41(10):2823-2831. doi: 10.1007/s00345-023-04549-y. Epub 2023 Aug 16. PMID 37587366
- [Background] Luo D, Wan X, Liu J, Tong T. Optimally estimating the sample mean from the sample size, median, mid-range, and/or mid-quartile range. Stat Methods Med Res. 2018 Jun;27(6):1785-1805. doi: 10.1177/0962280216669183. Epub 2016 Sep 27. PMID 27683581
- [Background] Kraft L, Yilmaz M, Petzold R, Gratzke C, Suarez-Ibarrola R, Miernik A. Dusting Efficiency of a Novel Pulsed Thulium:Yttrium Aluminum Garnet Laser vs a Thulium Fiber Laser. J Endourol. 2022 Feb;36(2):259-265. doi: 10.1089/end.2021.0441. Epub 2021 Nov 16. PMID 34693738
- [Background] Kraft L, Petzold R, Suarez-Ibarrola R, Miernik A. In vitro fragmentation performance of a novel, pulsed Thulium solid-state laser compared to a Thulium fibre laser and standard Ho:YAG laser. Lasers Med Sci. 2022 Apr;37(3):2071-2078. doi: 10.1007/s10103-021-03495-8. Epub 2021 Dec 14. PMID 34905141
- [Background] Korolev D, Akopyan G, Tsarichenko D, Shpikina A, Ali S, Chinenov D, Corrales M, Taratkin M, Traxer O, Enikeev D. Minimally invasive percutaneous nephrolithotomy with SuperPulsed Thulium-fiber laser. Urolithiasis. 2021 Oct;49(5):485-491. doi: 10.1007/s00240-021-01258-2. Epub 2021 Mar 3. PMID 33655346
- [Background] Huusmann S, Lafos M, Meyenburg I, Muschter R, Teichmann HO, Herrmann T. Tissue effects of a newly developed diode pumped pulsed Thulium:YAG laser compared to continuous wave Thulium:YAG and pulsed Holmium:YAG laser. World J Urol. 2021 Sep;39(9):3503-3508. doi: 10.1007/s00345-021-03634-4. Epub 2021 Mar 16. PMID 33728503
- [Background] Haas CR, Knoedler MA, Li S, Gralnek DR, Best SL, Penniston KL, Nakada SY. Pulse-modulated Holmium:YAG Laser vs the Thulium Fiber Laser for Renal and Ureteral Stones: A Single-center Prospective Randomized Clinical Trial. J Urol. 2023 Feb;209(2):374-383. doi: 10.1097/JU.0000000000003050. Epub 2023 Jan 9. PMID 36621994
- [Background] Flight L, Julious SA. Practical guide to sample size calculations: non-inferiority and equivalence trials. Pharm Stat. 2016 Jan-Feb;15(1):80-9. doi: 10.1002/pst.1716. Epub 2015 Nov 25. PMID 26604186
- [Background] Enikeev D, Grigoryan V, Fokin I, Morozov A, Taratkin M, Klimov R, Kozlov V, Gabdullina S, Glybochko P. Endoscopic lithotripsy with a SuperPulsed thulium-fiber laser for ureteral stones: A single-center experience. Int J Urol. 2021 Mar;28(3):261-265. doi: 10.1111/iju.14443. Epub 2020 Nov 30. PMID 33258271
- [Background] Corrales M, Traxer O. Retrograde intrarenal surgery: laser showdown (Ho:YAG vs thulium fiber laser). Curr Opin Urol. 2022 Mar 1;32(2):179-184. doi: 10.1097/MOU.0000000000000971. PMID 35013078
- [Background] Bergmann J, Rosenbaum CM, Netsch C, Gross AJ, Becker B. First Clinical Experience of a Novel Pulsed Solid-State Thulium:YAG Laser during Percutaneous Nephrolithotomy. J Clin Med. 2023 Mar 29;12(7):2588. doi: 10.3390/jcm12072588. PMID 37048670
- [Background] Azilgareeva, C., Taratkin, M., Petov, V., Korolev, D., Akopyan, G., Dymov, A., et al. (2022). Prospective randomized comparison of SP TFL and Ho:YAG in RIRS for kidney stones: a single-center study. Eur. Urol. 81, S1722-S1723. doi: 10.1016/S0302-2838(22)01252-0.
- [Background] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART I. J Urol. 2016 Oct;196(4):1153-60. doi: 10.1016/j.juro.2016.05.090. Epub 2016 May 27. PMID 27238616

DOCUMENTS (2):
  • Study Protocol (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT06721975/Prot_000.pdf
  • Informed Consent Form (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT06721975/ICF_001.pdf